CLINICAL TRIAL: NCT04248829
Title: A Phase III, Randomized, Double-blind Study to Assess the Efficacy and Safety of Lazertinib Versus Gefitinib as the First-line Treatment in Patients With Epidermal Growth Factor Receptor Sensitizing Mutation Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Clinical Trial of YH25448(Lazertinib) as the First-line Treatment in Patients With EGFR Mutation Positive Locally Advanced or Metastatic NSCLC (LASER301)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YH25448-301
Record Dates: First submitted 2020-01-14; First posted 2020-01-30 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Locally Advanced EGFR Sensitizing Mutation; Metastatic EGFR Sensitizing Mutation; EGFR TKI; Ex19del; L858R; First-line; YH25448; Advanced Non-Small Cell Lung Cancer; Adenocarcinoma of lung; Non-squamous carcinoma of lung; Phase III; Lazertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — lazertinib; Gefitinib

STUDY DESIGN:
Intervention Model Description: Approximately 380 patients will be randomized in a 1:1 ratio to either lazertinib (n=190) or gefitinib (n= 190).
  Following objective disease progression according to RECIST v1.1, as per investigator assessment, patients who were randomized to gefitinib arm may have the option to receive open-label lazertinib
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lazertinib + Gefitinib-matching placebo (Experimental): Lazertinib (240 mg or 160 mg orally, once daily) plus Gefitinib-matching placebo (250 mg orally, once daily) in accordance with the randomization schedule
  Interventions: Drug: Lazertinib 240 mg/160 mg; Drug: Gefitinib-matching placebo 250 mg
- Gefitinib + Lazertinib-matching placebo (Active Comparator): Gefitinib (250 mg orally, once daily) plus Lazertinib-matching placebo (240 mg or 160 mg orally, once daily) in accordance with the randomization schedule
  Interventions: Drug: Gefitinib 250 mg; Drug: Lazertinib-matching placebo 240 mg/160 mg

INTERVENTIONS:
Drug: Lazertinib 240 mg/160 mg — The initial dose of lazertinib 240 mg (3 tablets of 80 mg lazertinib) once daily can be reduced to 160 mg once daily (2 tablets of 80 mg lazertinib) under specific circumstances
  Other Names: YH25448 240 mg/160 mg
  Arms: Lazertinib + Gefitinib-matching placebo
Drug: Gefitinib 250 mg — The initial dose for Gefitinib (250 mg once daily) cannot be reduced to a lower dose
  Other Names: Iressa 250 mg
  Arms: Gefitinib + Lazertinib-matching placebo
Drug: Lazertinib-matching placebo 240 mg/160 mg — The initial dose of lazertinib-matching placebo 240 mg (3 tablets of 80 mg lazertinib-matching placebo) once daily can be reduced to 160 mg once daily (2 tablets of 80 mg lazertinib-matching placebo) under specific circumstances
  Other Names: YH25448-matching placebo 240 mg/160 mg
  Arms: Gefitinib + Lazertinib-matching placebo
Drug: Gefitinib-matching placebo 250 mg — The initial dose for Gefitinib-matching placebo (250 mg once daily) cannot be reduced to a lower dose
  Other Names: Iressa-matching placebo 250 mg
  Arms: Lazertinib + Gefitinib-matching placebo

SUMMARY:
This Phase III study will be conducted to evaluate the efficacy and safety of YH25448 as first-line treatment in locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) patients with EGFR mutations

DETAILED DESCRIPTION:
YH25448 is an oral, highly potent, mutant-selective and irreversible EGFR Tyrosine-kinase inhibitors (TKIs) that targets both the T790M mutation and activating EGFR mutations while sparing wild type EGFR.

This is a Phase III, Randomized, Double-blind study evaluating the efficacy and safety of YH25448 (240 mg orally, once daily) versus Gefitinib (250 mg orally, once daily) in patients with locally advanced or metastatic NSCLC that is known to be EGFR sensitizing mutation (EGFRm) positive, treatment-naïve and eligible for first-line treatment with an EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the lung
* Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy
* At least 1 of the 2 common EGFR mutations known to be associated with EGFR TKI sensitivity (Ex19del or L858R), either alone or in combination with other EGFR mutations
* Treatment-naïve for locally advanced or metastatic NSCLC
* WHO performance status score of 0 to 1 with no clinically significant deterioration over the previous 2 weeks before randomization
* At least 1 measurable lesion, not previously irradiated and not chosen for biopsy during the study Screening period

Exclusion Criteria:

* Symptomatic and unstable brain metastases
* Leptomeningeal metastases
* Symptomatic spinal cord compression
* History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD
* Any medical conditions requiring chronic continuous oxygen therapy
* History of any malignancy other than the disease under study within 3 years before randomization
* Any cardiovascular disease as follows:

  * History of symptomatic chronic heart failure or serious cardiac arrhythmia requiring active treatment
  * History of myocardial infarction or unstable angina within 24 weeks of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (80):
- Princess Alexandra Hospital, Woolloongabba, Queensland, Australia
- Greece (3):
  - Eugenideio Therapeutirio - Ongcology Department, Athens
  - Attikon Hospital, Athens
  - Theageneio Anticancer Hospital of Thessaloniki, Thessaloniki
- Hungary (2):
  - Debreceni Egyetem, Debrecen
  - Törökbálinti Tüdőgyógyintézet, Törökbálint
- Malaysia (6):
  - Hospital Sultan Ismail, Johor Bahru, Johor
  - Hospital Raja Perempuan Zainab Ii, Kota Bharu, Kelantan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Umum Sarawak, Kuching, Sarawak
  - University Malaya Medical Centre, Kuala Lumpur, Selangor
- Philippines (3):
  - Manila Doctors Hospital - Clinical Trial Office, Manila, Quezon
  - Perpetual Succour Hospital, Cebu
  - Philippine General Hospital, Manila
- Russia (15):
  - Arkhangelsk Regional Clinical Oncological Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - GBUZ of Nizhny Novgorod region Clinical diagnostic center, Nizhny Novgorod, Nizhny Novgorod Oblast
  - GAUZ Republican clinical oncology dispensary of the Ministry, Kazan'
  - Republic Clinical Oncology Despensary, Kazan'
  - Medincentre (GLAVUPDK), Moscow
  - VitaMed LLC, Moscow
  - MBUZ City Clinical Hospital #1, Novosibirsk
  - Budgetary Healthcare Institution of Omsk Region "Clinical Oncology Dispensary", Omsk
  - Private medical institution "Euromedservice", Pushkin
  - First St. Petersburg State Medical University n. a. Pavlov, Saint Petersburg
  - LLC "Eurocityclinic", Saint Petersburg
  - Limited Liability Company "AV Medical Group" - Oncology, Saint Petersburg
  - Saint-Petersburg City Clinical Oncology Dispensary, Saint Petersburg
  - GBUZ "Regional clinical oncologic dispensary of Volgograd", Volgograd
  - Yaroslavl regional oncology hospital, Yaroslavl
- Serbia (3):
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz, Vojvodina
  - Clinical Hospital Center "Bezanijska Kosa", Belgrade
  - Clinical Center Kragujevac, Kragujevac
- National University Hospital, Singapore, Singapore
- South Korea (22):
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St.Mary's Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (5):
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University - Faculty of Medicine, Chiang Mai
  - Prince of Songkla University, Hat Yai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
- Turkey (Türkiye) (9):
  - Adana Baskent Practice and Research Hospital, Adana
  - Cukurova University Medical Faculty, Adana
  - Ankara Liv Hospital, Ankara
  - Hacettepe University Medical Faculty - Medical Oncology, Ankara
  - Trakya University Medical Faculty, Edirne
  - Istanbul Medeniyet University Goztepe Training and Research Hospital - Medical Oncology, Istanbul
  - Medical Point İzmir Hospital, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Inonu University Turgut Ozal Medical Center, Malatya
- Ukraine (8):
  - Komunalne nekomertsiine pidpryiemstvo Kharkivskoi oblasnoi rady "Oblasnyi klinichnyi spetsializovanyi dyspanser radiatsiinoho zakhystu naselennia" - khirurhichne viddilennia, Kharkiv, Kharkivs’ka Oblast’
  - Tsentralna miska klinichna likarnia, Uzhhorod, Zakarpattia Oblast
  - Oblasne komunalne nekomertsiine pidpryiemstvo "Bukovynskyi klinichnyi onkolohichnyi tsentr", strukturnyi pidrozdil klinichnoi onkolohii, m.Chernivtsi, Chernivtsi
  - Komunalne nekomertsiine pidpryiemstvo "Miska klinichna likarnia №4" Dniprovskoi miskoi rady", khimioterapevtychne viddilennia z dennym statsionarom, Derzhavnyi zaklad "Dnipropetrovskyi derzhavnyi medychnyi universitet", kafedra onkolohii i medychnoi radio, Dnipro
  - Kyiv City Clinical Oncology Center - Department of Chemotherapy, Kyiv
  - Komunalne nekomertsiine pidpryiemstvo Sumskoi oblasnoi rady "Sumskyi klinichnyi onkolohichnyi tsentr", onkotorakalne viddilennia, Sumskyi derzhavnyi universytet, kafedra onkolohii ta radiolohii, m. Sumy, Sumy
  - Podilskyi rehionalnyi tsentr onkolohii, viddilennia khimioterapii, Vinnytsia
  - Medychnyi tsentr Tovarystva z obmezhenoiu vidpovidalnistiu "Onkolaif", Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underline the results reported in study-related publications will be made available during the period beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed. Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to hmbyun@yuhan.co.kr.
  Other documents(i.e. a summary of the study results, study protocol, statistical analysis plan) will be posted in the publicly accessible database (i.e. clinicaltrials.gov) no later than 1 year after the study's primary completion date.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed.
Access Criteria: Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to hmbyun@yuhan.co.kr.

REFERENCES:
- [Derived] Soo RA, Cho BC, Kim JH, Ahn MJ, Lee KH, Zimina A, Orlov S, Bondarenko I, Lee YG, Lim YN, Lee SS, Lee KH, Pang YK, Fong CH, Kang JH, Lim CS, Danchaivijitr P, Kilickap S, Yang JC, Arslan C, Lee H, Park SN, Cicin I. Central Nervous System Outcomes of Lazertinib Versus Gefitinib in EGFR-Mutated Advanced NSCLC: A LASER301 Subset Analysis. J Thorac Oncol. 2023 Dec;18(12):1756-1766. doi: 10.1016/j.jtho.2023.08.017. Epub 2023 Oct 22. PMID 37865896
- [Derived] Cho BC, Ahn MJ, Kang JH, Soo RA, Reungwetwattana T, Yang JC, Cicin I, Kim DW, Wu YL, Lu S, Lee KH, Pang YK, Zimina A, Fong CH, Poddubskaya E, Sezer A, How SH, Danchaivijitr P, Kim Y, Lim Y, An T, Lee H, Byun HM, Zaric B. Lazertinib Versus Gefitinib as First-Line Treatment in Patients With EGFR-Mutated Advanced Non-Small-Cell Lung Cancer: Results From LASER301. J Clin Oncol. 2023 Sep 10;41(26):4208-4217. doi: 10.1200/JCO.23.00515. Epub 2023 Jun 28. PMID 37379502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 393 participants were randomized to treatment at 96 study sites in 13 countries.
Pre-assignment Details: During the 28 day screening period, participants were enrolled based on the presence in their tumour of at least 1 of the 2 most frequent Epidermal growth factor receptor (EGFR) mutations. At the time of enrolment, all participants were required to provide biopsy tissue for central testing of the Exon 19 deletion (Ex19del) and L858R mutations.
Groups:
- Lazertinib 240 mg: Randomized participants received Lazertinib 240 mg orally once daily (QD)
- Gefitnib 250 mg: Randomized participants received Gefitinib 250 mg orally once daily (QD)
Period: Overall Study
Arm/Group | Lazertinib 240 mg | Gefitnib 250 mg
Started | 196 | 197
Completed (Participants ongoing study treatment at data cut-off) | 108 | 47
Not Completed | 88 | 150
Not completed — Disease progression | 44 | 109
Not completed — Adverse Event | 19 | 18
Not completed — Withdrawal by Subject | 11 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 12 | 14
Not completed — Physician Decision | 2 | 4
Not completed — Any reason not specifically recorded | 0 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS), FAS included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lazertinib 240 mg | Gefitnib 250 mg | Total
Number analyzed (Participants) | 196 | 197 | 393
Age, Customized [Median (Full Range); unit: years] | 67 [31 to 87] | 64 [25 to 86] | 65 [25 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 119 | 251
  Male | 64 | 78 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 130 | 130 | 260
  Race: Non-Asian | 66 | 67 | 133
Smoking history [Count of Participants; unit: Participants]
  Never | 135 | 149 | 284
  Former | 50 | 42 | 92
  Current | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) According to RECIST v1.1 by Investigator Assessment
Description: PFS was defined as the time from randomization until the date of objective progression or death(by any cause whichever comes first based on investigator assessment using RECIST v1.1 and was used to assess the efficacy of lazertinib compared to the gefitinib).
Time Frame: At baseline and every 6 weeks for the first 18 months and then every 12 weeks relative to randomization until progression, assessed up to 29 months per participant.
Population: The full analysis set (FAS), FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lazertinib 240 mg | Gefitnib 250 mg
Number analyzed (Participants) | 196 | 197
Months | 20.6 [17.8 to 26.1] | 9.7 [9.2 to 11.3]

2. Secondary Outcome: Objective Response Rate (ORR) According to RECIST v1.1 by Investigator Assessments
Description: ORR was defined as the percentage of participants with measurable disease with at least on visit response of complete response(CR) or Partial response(PR) and it was used to further assess the efficacy of lazertinib compared with gefitinib.
Time Frame: as for outcome 1
Population: The full analysis set (FAS), FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lazertinib 240 mg | Gefitnib 250 mg
Number analyzed (Participants) | 196 | 197
Percentage of participants | 76.0 [69.4 to 81.8] | 76.1 [69.6 to 81.9]

3. Secondary Outcome: Duration of Response (DoR) According to RECIST v1.1 by Investigator Assessments
Description: DoR was defined as the time from the date of first documented response(CR or PR) until the date of documented progression or death, whichever comes first and was used to further assess the efficacy of lazertinib compared with gefitinib.
Time Frame: as for outcome 1
Population: The full analysis set (FAS), FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lazertinib 240 mg | Gefitnib 250 mg
Number analyzed (Participants) | 196 | 197
Months | 19.4 [16.6 to 24.9] | 8.3 [6.9 to 10.9]

4. Secondary Outcome: Disease Control Rate (DCR) According to RECIST v1.1 by Investigator Assessments
Description: DCR was defined as the percentage of participants who have a best overall response of CR or PR or SD(SD at >= 6weeks prior to any PD event) and was used to further assess the efficacy of lazertinib compared with gefitinib.
Time Frame: as for outcome 1
Population: The full analysis set (FAS), FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lazertinib 240 mg | Gefitnib 250 mg
Number analyzed (Participants) | 196 | 197
Percentage of participants | 93.9 [89.5 to 96.8] | 93.9 [89.6 to 96.8]

5. Secondary Outcome: Depth of Response According to RECIST v1.1 by Investigator Assessments
Description: The depth of response was defined as the best percent change in the sum of diameters of target lesions in the absense of new lesions or progression of non-target lesions compared to the baseline and was used to further assess the efficacy of lazertinib compared with gefitinib.
Time Frame: At baseline and every 6 weeks for the first 18 months and then every 12 weeks relative to randomization until progression.
Reporting Status: Not Posted

6. Secondary Outcome: Time to Response According to RECIST v1.1 by Investigator Assessments
Description: Time to Response was defined as the time from the date of randomization until the date of first documented response and was used to further assess the efficacy of lazertinib compared with gefitinib.
Time Frame: as for outcome 5
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death due to any cause and was used to further assess the efficacy of lazertinib compared with gefitinib.
Time Frame: From the randomization to end of study or date of death from any cause, whichever comes first, assessed every 6 weeks. (Up to 29 months per participant.)
Population: The full analysis set (FAS), FAS included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Lazertinib 240 mg | Gefitnib 250 mg
Number analyzed (Participants) | 196 | 197
Participants
  Death | 49 | 64
  Alive/Censored | 147 | 133

8. Secondary Outcome: Plasma Concentrations of Lazertinib
Description: To characterize the pharmacokinetics (PK) of lazertinib.
Time Frame: Blood samples collected from each participant at pre-dose, 1 to 3 hours, and 4 to 6 hours post-dose on Day 1 Cycle 1, Day 1 Cycle 2, Day 1 Cycle 5, Day 1 Cycle 9, and Day 1 Cycle 13.
Reporting Status: Not Posted

9. Secondary Outcome: Cerebrospinal Fluid (CSF) Concentrations of Lazertinib
Description: To characterize the pharmacokinetics (PK) of lazertinib.
Time Frame: A cerebrospinal fluid (CSF) sample once collected from participants with brain metastases, at Cycle 5 Day 1 or afterward.
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 Items (QLQ-C30)
Description: The EORTC QLQ-C30 consists of 30 items and measures cancer participants' functioning (health related quality of life (HRQoL)) and symptoms for all cancer types. Questions can be grouped into 5 multi item functional scales (physical, role, emotional, cognitive, and social); 3 multi item symptom scales (fatigue, pain, nausea/vomiting); a 2 item global HRQoL scale; 5 single items assessing additional symptoms commonly reported by cancer participants (dyspnea, loss of appetite, insomnia, constipation, diarrhea) and 1 item on the financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  * a high score for a functional scale represents a high / healthy level of functioning
  * a high score for the global health status / QoL represents a high QoL
  * but a high score for a symptom scale / item represents a high level of symptomatology / problems
Time Frame: Questionnaires completed at Cycle 1 Day1 , Cycle2 Day 1 and then every 6 weeks relative to the randomization date until 28d safety f/u or progression f/u visit(whichever is later).
Reporting Status: Not Posted

11. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Lung Cancer 13 Items (EORTC QLQ-LC13)
Description: The EORTC QLQ-LC13 includes questions assessing cough, hemoptysis, dyspnea, site specific pain (symptoms), sore mouth, dysphagia, peripheral neuropathy, and alopecia (treatment related side effects), and pain medication.
  The items on both measures were scaled and scored using the recommended EORTC procedures. Raw scores were transformed to a linear scale ranging from 0 to 100, with a higher score representing a higher level of functioning or higher level of symptoms. Provided at least half of the items in the scale were completed, the scale score was calculated using only those items for which values existed.
Time Frame: as for outcome 10
Reporting Status: Not Posted

12. Secondary Outcome: Change From Baseline in Euro-Quality of Life-5 Dimension-5 Level (EQ-5D-5L)
Description: The EQ-5D comprises the following two questionnaires:
  * The EQ-5D comprises 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension comprises five levels (no problems, slight problems, moderate problem, severe problem, unable/extreme problems).
  * The EQ VAS records the participants self-rated health status on a vertical graduated (0-100) visual analogue scale. The patient's self-rated health is assessed on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state) by the EQ-VAS.
Time Frame: as for outcome 10
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from the time of signature of informed consent throughout the Treatment Period and including the safety follow-up period.The safety follow-up period was defined as 28 days after study drug was discontinued. (Up to 29 months per participant.)
Description: An adverse event was the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. In clinical studies, an AE included an undesirable medical condition occurring at any time, even if no study treatment had been administered. The term AE was used to include both serious and non-serious AEs.
Arm/Group | Lazertinib 240 mg | Gefitnib 250 mg
All-Cause Mortality (participants affected / at risk) | 49/196 | 64/197
Serious Adverse Events (participants affected / at risk) | 51/196 | 51/197
Other Adverse Events (participants affected / at risk) | 189/196 | 188/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lazertinib 240 mg (N=196) | Gefitnib 250 mg (N=197)
COVID-19 (Infections and infestations) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 8 | 3
Actinomycosis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 3
Bronchitis (Infections and infestations) | 0 | 2
Infectious pleural effusion (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Death (General disorders) | 3 | 3
Oedema peripheral (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 4
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lazertinib 240 mg (N=196) | Gefitnib 250 mg (N=197)
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 19
Rash (Skin and subcutaneous tissue disorders) | 71 | 72
Pruritus (Skin and subcutaneous tissue disorders) | 52 | 36
Paronychia (Skin and subcutaneous tissue disorders) | 35 | 34
Dry skin (Skin and subcutaneous tissue disorders) | 29 | 23
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 21 | 27
Paraesthesia (Nervous system disorders) | 77 | 13
Headache (Nervous system disorders) | 18 | 10
Dizziness (Nervous system disorders) | 11 | 10
Diarrhoea (Gastrointestinal disorders) | 51 | 77
Stomatitis (Gastrointestinal disorders) | 31 | 16
Nausea (Gastrointestinal disorders) | 30 | 18
Constipation (Gastrointestinal disorders) | 28 | 20
Vomiting (Gastrointestinal disorders) | 10 | 14
Alanine aminotransferase increased (Investigations) | 30 | 59
Aspartate aminotransferase increased (Investigations) | 22 | 52
Blood alkaline phosphatase increased (Investigations) | 12 | 12
Weight decreased (Investigations) | 9 | 14
Gamma-glutamyltransferase increased (Investigations) | 8 | 13
COVID-19 (Infections and infestations) | 16 | 14
Urinary tract infection (Infections and infestations) | 10 | 14
Pneumonia (Infections and infestations) | 10 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 14
Decreased appetite (Metabolism and nutrition disorders) | 33 | 31
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 8
Fatigue (General disorders) | 16 | 8
Asthenia (General disorders) | 12 | 8
Anaemia (Blood and lymphatic system disorders) | 36 | 23
Insomnia (Psychiatric disorders) | 11 | 11
thrombocytopenia (Blood and lymphatic system disorders) | 13 | 7
Hypertension (Vascular disorders) | 8 | 10
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Dyspepsia (Gastrointestinal disorders) | 10 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 3
Oedema peripheral (General disorders) | 12 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT04248829/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT04248829/SAP_001.pdf